CLINICAL TRIAL: NCT03797014
Title: Efficacy, Safety, and Tolerability of Bictegravir/Emtricitabine/Tenofovir Alafenamide in Adults With HIV-HBV Coinfection
Brief Title: B/F/TAF Switch Study for HIV-HBV Coinfection
Acronym: BEST-HBV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Joel Chua, Assistant Professor of Medicine, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP00083844
Record Dates: First submitted 2019-01-04; First posted 2019-01-08 (Actual); Results first posted 2023-07-18 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: HIV-1-infection; Hepatitis B
Keywords: HIV-1; Hepatitis B; HIV-HBV coinfection; Bictegravir; B/F/TAF; Tenofovir alafenamide; Biktarvy
MeSH Terms: conditions — Hepatitis B | interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Intervention Model Description: This is an open-label phase 4 switch study to evaluate the efficacy, safety, and tolerability of FDC B/F/TAF in adults with HIV-1 and HBV coinfection.
Masking Description: This is an open label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- B/F/TAF (Experimental): Treatment group (1-arm study)
  Interventions: Drug: B/F/TAF

INTERVENTIONS:
Drug: B/F/TAF — Fixed dose combination B/F/TAF (50 mg/ 200 mg/ 25 mg/ tablet) administered orally once daily without regards to food.
  Other Names: Bictegravir/emtricitabine/tenofovir alafenamide

SUMMARY:
The primary objective of this study is to evaluate the efficacy and safety of fixed dose combination (FDC) bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) in adults coinfected with both HIV-1 and hepatitis B. As this is a switch study, all eligible subjects enrolled will be switched from their current antiretroviral regimen to B/F/TAF will be followed on treatment for 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older at enrollment.
2. Documented HIV-1 infection and currently on a stable regimen for at least 3 months if on an INSTI-based regimen (6 months if on a non-INSTI-based regimen) preceding the screening visit with documented plasma HIV-1 RNA ≤ 50 copies/mL for at least 3 months preceding the screening visit.
3. No known history of resistance to tenofovir alafenamide (TAF), emtricitabine (FTC), or Bictegravir (BIC).
4. Documented chronic hepatitis B infection, based on any of the following: a. Positive HBsAg result or nucleic acid test for HBV DNA (including qualitative, quantitative, and genotype testing) or positive HBeAg on two occasions at least 6 months apart (any combination of these tests performed 6 months apart is acceptable); or b. Negative immunoglobulin M (IgM) antibodies to HBV core antigen (anti-HBc IgM) AND a positive results on one of the following tests: HBsAg, HBeAg, or nucleic acid test for HBV DNA (including qualitative, quantitative, and genotype testing) prior to or at screening.
5. No current or prior regimen containing three active anti-HBV agents (i.e. cannot be on tenofovir alafenamide (TDF)/emtricitabine (FTC)/entecavir or TDF/lamivudine (3TC)/entecavir).
6. Must have a primary care provider(s) for medical management.
7. Females of childbearing potential must agree to utilize protocol recommended highly effective contraceptive methods or be non-heterosexually active or practice sexual abstinence from screening and throughout the duration of the study. Female subjects who utilize hormonal contraceptive as one of their birth control methods must have used the same method for at least 3 months prior to study drug dosing.
8. Male subjects must be willing to abstain from heterosexual intercourse or use a condom throughout the study period.
9. Stated willingness to comply with all study procedures and availability for the duration of the study.
10. Written informed consent must be obtained before any study procedure is performed.

Exclusion Criteria:

1. Females who are pregnant or breastfeeding.
2. Any known allergies to any of the components of B/F/TAF.
3. Treatment with another investigational drug within three months of enrollment.
4. Abnormal hematological and biochemical parameters at screening, including:

   1. Absolute neutrophil count (ANC) < 750 cells/mm3.
   2. Platelets < 50,000/mm3.
   3. Hemoglobin < 8.5 g/dL.
   4. AST or ALT of > 5 times upper limit of normal (ULN).
   5. Estimated GFR < 30 mL/min/1.73 m2.
   6. Total bilirubin > 1.5 times ULN.
5. Previous or current history of malignancy, other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, non-invasive cutaneous squamous cell carcinoma. Note: Those with a history of malignancy who are in remission for two or more years may be included in the study.
6. An opportunistic illness indicative of stage 3 HIV diagnosed within the 30 days prior to screening.
7. Subjects experiencing decompensated cirrhosis (e.g. ascites, encephalopathy, or variceal bleeding).
8. Acute hepatitis in the 30 days prior to study entry.
9. Active tuberculosis infection.
10. Subjects receiving ongoing therapy with any medications contraindicated for co-administration with B/F/TAF FDC, including but not limited to the following medications: dofetilide, phenobarbital, phenytoin, carbamazepine, oxcarbamazepine, rifampin, rifapentine, cisapride, St. John's Wort, and Echinaceae.
11. Current alcohol or substance use that in the opinion of the investigator may interfere with subject study compliance.
12. Any other clinical conditions that in the opinion of the investigator would make the subject unsuitable for the study or unable to comply with the dosing requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2023-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel V Chua, MD, Principal Investigator — Institute of Human Virology, University of Maryland
Locations (2):
- United States (2):
  - Institute of Human Virology Clinical Research Unit, Baltimore, Maryland
  - Newlands Health, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Individual participant data is available upon reasonable request from the investigator.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | B/F/TAF
Started | 28
Completed | 25
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | B/F/TAF
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 3
Age, Continuous [Mean (Full Range); unit: years] | 50.1 [28 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 25
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 28
HIV RNA PCR <50 copies/mL [Count of Participants; unit: Participants] | 20
CD4 count <200 cells/microliter [Count of Participants; unit: Participants] | 1
HBV DNA PCR <29 IU/mL [Count of Participants; unit: Participants] | 22
HBeAg positive [Count of Participants; unit: Participants] | 12
Anti-HBe antibody positive [Count of Participants; unit: Participants] | 10
Abnormal ALT [Count of Participants; unit: Participants] | 4
Hepatitis D antibody positive [Count of Participants; unit: Participants] | 5

OUTCOME MEASURES:

1. Primary Outcome: HIV-1 RNA at Week 24
Description: Proportion of participants with HIV-1 RNA <50 copies/mL at Week 24 by US FDA Snapshot Algorithm
Time Frame: Week 24
Population: Intention-to-Treat (ITT) population: Enrolled subjects who received at least one study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | B/F/TAF
Number analyzed (Participants) | 28
Participants | 25

2. Primary Outcome: HBV DNA at Week 24
Description: Proportion of participants with plasma HBV DNA <29 IU/mL at Week 24 as defined by Missing=Failure Approach
Time Frame: Week 24
Population: Intention-to-Treat Population: All enrolled subjects who received at least one study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | B/F/TAF
Number analyzed (Participants) | 28
Participants | 24

3. Secondary Outcome: HIV-1 RNA at Week 48
Description: Proportion of participants with HIV-1 RNA <50 copies/mL at Week 48 by US FDA Snapshot Algorithm
Time Frame: Week 48
Population: Intention-to-Treat Population: All enrolled subjects who received at least one study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | B/F/TAF
Number analyzed (Participants) | 28
Participants | 22

4. Secondary Outcome: HBV DNA at Week 48
Description: Proportion of participants with plasma HBV DNA <29 IU/mL at Week 48 as defined by Missing=Failure Approach
Time Frame: Week 48
Population: Intention-to-Treat Population: All enrolled subjects who received at least one study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | B/F/TAF
Number analyzed (Participants) | 28
Participants | 22

5. Secondary Outcome: CD4 Cell Count Change at Week 24
Description: Change from baseline in CD4 cell count at Week 24
Time Frame: Baseline; Week 24
Population: All enrolled subjects with CD4 count values at baseline and at week 24.
Measure: Mean (Standard Deviation); unit: cells/microliter
Arm/Group | B/F/TAF
Number analyzed (Participants) | 26
cells/microliter | 32.8 (169.1)

6. Secondary Outcome: CD4 Cell Count Change at Week 48
Description: Change from baseline in CD4 cell count at Week 48
Time Frame: Baseline; Week 48
Population: All enrolled subjects with CD4 count results available at baseline and week 48.
Measure: Mean (Standard Deviation); unit: cells/microliter
Arm/Group | B/F/TAF
Number analyzed (Participants) | 25
cells/microliter | 76.6 (184.2)

7. Secondary Outcome: ALT Normalization at Week 24
Description: Proportion of participants with normal ALT at Week 24
Time Frame: Week 24
Population: Enrolled subjects with abnormal ALT at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | B/F/TAF
Number analyzed (Participants) | 4
Participants | 4

8. Secondary Outcome: ALT Normalization at Week 48
Description: Proportion of participants with normal ALT at Week 48
Time Frame: Week 48
Population: All enrolled subjects with abnormal baseline LFTs
Measure: Count of Participants; unit: Participants
Arm/Group | B/F/TAF
Number analyzed (Participants) | 4
Participants | 4

9. Secondary Outcome: HBeAg Loss at Week 48
Description: Proportion of participants with hepatitis B envelop antigen (HBeAg) loss at Week 48 visit.
Time Frame: Week 48
Measure: Count of Participants; unit: Participants
Arm/Group | B/F/TAF
Number analyzed (Participants) | 26
Participants | 0

10. Secondary Outcome: HBsAg Loss at Week 48
Description: Proportion of participants with hepatitis B surface antigen (HBsAg) loss at Week 48 visit.
Time Frame: Week 48
Measure: Count of Participants; unit: Participants
Arm/Group | B/F/TAF
Number analyzed (Participants) | 25
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the entire study participation (48 weeks).
Description: Adverse events were graded according to the Division of AIDS (DIADS) Table for Grading the Severity of Adult and Pediatric Adverse Events, version 2.1 (March 2017).
Arm/Group | B/F/TAF
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 16/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | B/F/TAF (N=28)
Upper respiratory tract infection (Infections and infestations) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Abscess, extremity (Infections and infestations) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (2)
Hypertension (Vascular disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
This study did not achieve its enrollment target of 60 and was adversely affected by COVID-19 pandemic travel and research restrictions particularly during April 2020 to August 2020.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-16): https://cdn.clinicaltrials.gov/large-docs/14/NCT03797014/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-31): https://cdn.clinicaltrials.gov/large-docs/14/NCT03797014/ICF_001.pdf